CLINICAL TRIAL: NCT03944213
Title: Resting-state Functional Connectivity Throughout a Course of iTBS in Major Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Clemens Mielacher, University Hospital, Bonn (Unknown); Maximilian Kiebs, University Hospital, Bonn (Unknown)
Responsible Party: Principal Investigator, Rene Hurlemann, Chair of the Medical Psychology Division and Deputy Chair of the Department of Psychiatry, University Hospital, Bonn
Other Study IDs: DepRest
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Depression; Depressive Disorder; Depressive Disorder, Major; Depressive Episode
Keywords: Transcranial Magnetic Stimulation; Theta Burst Stimulation; rTMS; TBS; resting-state fMRI
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD patients
  Interventions: Device: intermittent theta burst stimulation (iTBS)
- Healthy controls

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) — 20 sessions of iTBS
  Groups: MDD patients

SUMMARY:
This study aims to investigate changes in functional connectivity over a four week treatment course with intermittent theta burst stimulation (iTBS) in patients with major depressive disorder (MDD). To this end, seven weekly resting-state fMRI (rs-fMRI) scans at 7 tesla (7T) will precede, accompany and follow the iTBS treatment course. By obtaining several samples of the modulatory effects of iTBS on functional connectivity networks and simultaneous measurements of the depressive symptoms it will be possible to assess the time course of changes in connectivity across different networks, and to assess the overall relationship between the network modulation and the antidepressant effects of the treatment over time.

DETAILED DESCRIPTION:
The immense disease burden of major depressive disorder (MDD) and unsatisfactory response rates to pharmacological and psychological interventions highlight the need for further development of treatment alternatives. The development of these alternatives relies on an understanding of the pathophysiology of depression, which has, despite considerable efforts, remained largely elusive. Findings have converged on the proposition that depression cannot be attributed to a singular factor and is better understood as a dysfunctional interaction of multiple parameters. At the neural level, depression is described as a dysfunction of several cortical and sub-cortical networks associated with affective salience, cognitive control and self-reverential thoughts. Encouragingly, several studies have shown that pathological alterations in one of these networks, the Default Mode network, may normalize following several weeks of treatment using repetitive transcranial magnetic stimulation (rTMS), an accepted treatment for major depression.

The present study aims to elucidate the time course of this modulatory effect on the different networks showing pathological connectivity profiles. Specifically, our aim is to obtain several measurements of functional connectivity and concomitant measures of the symptoms of depression prior to, throughout, and following the 4 week treatment course of iTBS, a faster but equally effective non-invasive brain stimulation technique compared to rTMS. Due to the fact that weekly changes in network connectivity are expected to be relatively small, the stronger BOLD Signal at 7T and the fact that peak temporal correlation coefficients calculated between network nodes have been shown to be significantly higher at 7T than 3T (e.g.) in the Default Mode network should greatly aid in detecting these differences. At each of the 7 measurement time points, fluctuations of BOLD signal will be recorded during a rs-fMRI scan lasting about 15 minutes. Our approach will allow to characterize the temporal profiles of the antidepressant effects of iTBS, thereby furthering our understanding of the mechanism by which iTBS contributes to the normalization of pathological neural connectivity and the reduction of depression symptoms. This proposed longitudinal functional imaging of therapeutic changes is highly relevant to the field of clinical neuroscience and should further advance our understanding of the pathophysiology of depression.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to provide consent.
* Diagnosis of Major Depressive Disorder according to DSM-V criteria.
* The duration of the current episode is at least four weeks and no more than five years.
* During the current episode, at least one antidepressant (adequate duration and dosage) was not effective OR at least two antidepressants were intolerable due to side effects.

Exclusion Criteria:

* The participant does not fulfill requirements for iTBS treatment according to safety guidelines.
* Cardiac or neurological surgery, active implants, metal parts within the body, claustrophobia.
* Pregnancy or breast-feeding.
* Psychiatric illness, e.g. substance abuse, psychosis, bipolar disorder, anorexia, obsessive compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder, personality disorder.
* Antipsychotic medication not approved for the treatment of depression.
* Acute suicidality.
* Conditions related to increased intracranial pressure.
* Brain injury or stroke.
* History of epilepsy in patient or in first-degree relative.
* Cerebral aneurysm.
* Neurological illness (e.g. dementia (score of less than 25 in Mini Mental State Exam), Parkinson's disease, chorea huntington, multiple sclerosis).
* Course of electroconvulsive therapy (ECT) within the last three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Outpatients at the psychiatric hospital of the University Hospital Bonn. The patients diagnosis of major depressive disorder will be verified via the structured clinical interview for DSM-5. iTBS protocols in line with international standards administered by a trained professional.
  Additionally, a healthy control sample is included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in functional connectivity coefficients based on rs-fMRI over 7 timepoints. | Six weekly measurements starting 1 week before first iTBS treatment session, one follow-up measurement four weeks after last measurement.
  Seed-to-voxel functional connectivity analysis of rs-fMRI data.

SECONDARY OUTCOMES:
Change in depression severity as measured by the Hamilton Depression Rating Scale (HDRS-17) over 7 timepoints. | Six weekly measurements starting 1 week before first iTBS treatment session, one follow-up measurement four weeks after last measurement.
  Remission defined as HDRS-17 score (range: 0 to 52) of less than or equal to 8 after the iTBS course. Response defined as a reduction of at least 50% from baseline in HDRS-17 score after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: René Hurlemann, Prof., Principal Investigator — University Hospital, Bonn
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Souery D, Papakostas GI, Trivedi MH. Treatment-resistant depression. J Clin Psychiatry. 2006;67 Suppl 6:16-22. PMID 16848672
- [Background] Hasler G. Pathophysiology of depression: do we have any solid evidence of interest to clinicians? World Psychiatry. 2010 Oct;9(3):155-61. doi: 10.1002/j.2051-5545.2010.tb00298.x. PMID 20975857
- [Background] Kaiser RH, Andrews-Hanna JR, Wager TD, Pizzagalli DA. Large-Scale Network Dysfunction in Major Depressive Disorder: A Meta-analysis of Resting-State Functional Connectivity. JAMA Psychiatry. 2015 Jun;72(6):603-11. doi: 10.1001/jamapsychiatry.2015.0071. PMID 25785575
- [Background] Fischer AS, Keller CJ, Etkin A. The Clinical Applicability of Functional Connectivity in Depression: Pathways Toward More Targeted Intervention. Biol Psychiatry Cogn Neurosci Neuroimaging. 2016 May;1(3):262-270. doi: 10.1016/j.bpsc.2016.02.004. Epub 2016 Mar 2. PMID 29560882
- [Background] Liston C, Chen AC, Zebley BD, Drysdale AT, Gordon R, Leuchter B, Voss HU, Casey BJ, Etkin A, Dubin MJ. Default mode network mechanisms of transcranial magnetic stimulation in depression. Biol Psychiatry. 2014 Oct 1;76(7):517-26. doi: 10.1016/j.biopsych.2014.01.023. Epub 2014 Feb 5. PMID 24629537
- [Background] Philip NS, Barredo J, van 't Wout-Frank M, Tyrka AR, Price LH, Carpenter LL. Network Mechanisms of Clinical Response to Transcranial Magnetic Stimulation in Posttraumatic Stress Disorder and Major Depressive Disorder. Biol Psychiatry. 2018 Feb 1;83(3):263-272. doi: 10.1016/j.biopsych.2017.07.021. Epub 2017 Aug 8. PMID 28886760
- [Background] Berlim MT, van den Eynde F, Tovar-Perdomo S, Daskalakis ZJ. Response, remission and drop-out rates following high-frequency repetitive transcranial magnetic stimulation (rTMS) for treating major depression: a systematic review and meta-analysis of randomized, double-blind and sham-controlled trials. Psychol Med. 2014 Jan;44(2):225-39. doi: 10.1017/S0033291713000512. Epub 2013 Mar 18. PMID 23507264
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Hale JR, Brookes MJ, Hall EL, Zumer JM, Stevenson CM, Francis ST, Morris PG. Comparison of functional connectivity in default mode and sensorimotor networks at 3 and 7T. MAGMA. 2010 Dec;23(5-6):339-49. doi: 10.1007/s10334-010-0220-0. Epub 2010 Jul 13. PMID 20625794